16.1.9 Documentation of Statistical Methods



# STATISTICAL ANALYSIS PLAN

**Study Protocol Number:** 

E6011-J081-202

i (diliber.

**Study Protocol** 

Title:

A Phase 2 Study of E6011 in Subjects With Rheumatoid Arthritis

Inadequately Responding to Biologics

**Date:** 4 Jun2018

**Version:** Version 1.0

# 1 TABLE OF CONTENTS

| 1 | LABLE | OF CONTENTS | |
|---|---|---|---|
| 2 | | ABBREVIATIONS AND DEFINITIONS OF TERMS | |
| 3 | | UCTION | |
| | | dy Objectives | |
| | 3.1.1 | Primary Objectives | 8 |
| | 3.1.2 | Secondary Objective | |
| | 3.1.3 | Exploratory Objective | 8 |
| | 3.2 Ove | erall Study Design and Plan | 8 |
| 4 | DETERM | IINATION OF SAMPLE SIZE | 9 |
| 5 | STATIST | ICAL METHODS | 9 |
| | 5.1 Stu | dy Endpoints | 9 |
| | 5.1.1 | Primary Endpoint | 9 |
| | 5.1.2 | Secondary Endpoints | 10 |
| | 5.2 Stu | dy Subjects | 11 |
| | 5.2.1 | Definitions of Analysis Sets | 11 |
| | 5.2.2 | Subject Disposition | 12 |
| | 5.2.3 | Protocol Deviations | 12 |
| | 5.2.4 | Demographic and Other Baseline Characteristics | |
| | 5.2.5 | Prior and Concomitant Therapy | 15 |
| | <b>5.2.6</b> | Treatment Compliance | |
| | 5.3 Dat | a Analysis General Considerations | |
| | 5.3.1 | Pooling of Centers | |
| | 5.3.2 | Adjustments for Covariates | |
| | 5.3.3 | Multiple Comparisons/Multiplicity | |
| | 5.3.4 | Examination of Subgroups | |
| | 5.3.5 | Handling of Missing Data, Dropouts, and Outliers | |
| | 5.3.6 | Other Considerations | |
| | 5.3.<br>5.3. | $oldsymbol{J}$ | |
| | | cacy Analyses | |
| | 5.4.1 | Primary Efficacy Analyses | |
| | 5.4.2 | Secondary Efficacy Analyses | |
| | 5.4.3 | Other Efficacy Analyses | |
| | | rmacokinetic, Pharmacodynamic, Pharmacogenomic, and Other | 20 |
| | | marker Analyses | 20 |
| | 5.5.1 | Pharmacokinetic Analyses | |
| | Sen | um E6011 Concentration | |

| | 5.5.2 | Pharmacodynamic, Pharmacogenomic, and Other Biomarker<br>Analyses | 21 |
|---|---|---|---|
| | 5.5. | 2.1 Pharmacodynamic, Pharmacogenomic Analyses | |
| | 5.5. | ullet | |
| | 5.5. | 2.3 Immunogenicity Analyses | 22 |
| | 5.6 Safe | ety Analyses | 23 |
| | 5.6.1 | Extent of Exposure | 23 |
| | 5.6.2 | Adverse Events | 24 |
| | 5.6.3 | Laboratory Values | 26 |
| | 5.6.4 | Vital Signs | 26 |
| | 5.6.5 | <b>Electrocardiograms</b> | |
| | 5.6.6 | Other Safety Analyses | |
| | 5.6. | | |
| | | 6.2 Neurological findings | |
| | | er Analyses | |
| | 5.7.1 | | |
| | | oloratory Analyses | |
| | _ | ension Phase Analyses | |
| 6 | | I ANALYSES | |
| 7 | | S IN THE PLANNED ANALYSES | |
| 8 | | IONS AND CONVENTIONS FOR DATA HANDLING | |
| | | eline, Time Windows for statistical analyses | |
| | 8.1.1 | Definition of baseline value | |
| | 8.1.2 | Definition of change from baseline and percent change from | |
| | | baseline | 30 |
| | 8.1.3 | Time windows | 30 |
| | 8.2 Pha | rmacokinetic data handling | |
| | <b>8.2.1</b> | Lower Limit of Quantification of E6011 Serum Concentration | 32 |
| | 8.2.2 | BLQ Handling for Developing Concentration-Time Profiles | 33 |
| | 8.2.3 | BLQ Handling for Developing Tables | 33 |
| | 8.2.4 | Handling of anomalous concentration values | 33 |
| | 8.2.5 | General Rules for Presentation of Drug Concentrations | 33 |
| | 8.3 Imp | outation rule for partial date | 33 |
| | 8.3.1 | Date of Diagnosis | 33 |
| | 8.3.2 | Medication | 34 |
| | 8.3.3 | Adverse Events | 34 |
| | 8.4 Dec | simal places | 35 |
| | 8.5 TN | F Agent | 36 |

| 9 | PRO | GRAMMING SPECIFICATIONS | 36 |
|---|---|---|---|
| 10 | STA | TISTICAL SOFTWARE | 36 |
| 11 | MOC | CK TABLES, LISTINGS, AND GRAPHS | 36 |
| 12 | REF | ERENCES | 37 |
| 13 | APP | ENDICES | 38 |
| | 13.1 | National Institute for Health: Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | 38 |
| | 13.2 | Sponsor's Grading for Determining Markedly Abnormal Laboratory Results | 40 |

# 2 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Term |
|--------------|-------------------------------------------------|
| ACR | American College of Rheumatology |
| AE | adverse event |
| ATC | anatomical therapeutic class |
| ANCOVA | analysis of covariance |
| Ang2 | angiopoietin 2 |
| ATC | anatomical therapeutic class |
| BLQ | below the limit of quantification |
| BMI | body mass index |
| BP | Blood pressure |
| CCP | cyclic citrullinated peptide |
| CDAI | clinical disease activity index |
| CI | confidence interval |
| CRF | case report form |
| CRP | C-reative Protein |
| CSR | clinical study report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DAS28 | disease activity score in 28 joints, |
| DP | Decimal places |
| EGF | epidermal growth factor |
| ESR | Erythrocyte Sedimentation Rate |
| EULAR | European League Against Rheumatism |
| FAS | full analysis set |
| γ-GTP | γ-glutamine transpeptidase |
| HAQ | Health Assessment Questionnare |
| HAQ-DI | Health Assessment Questionnare Disability Index |
| IL | Interleukin |
| LLOQ | lower limit of quantification |
| LOCF | last observation carried forward |

Eisai 

| Abbreviation | Term |
|--------------|-------------------------------------------------------|
| LRG1 | leucine-rich alpha-2 glycoprotein 1 |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMP | matrix metalloproteinase |
| MTX | Methotrexate |
| NCI | National Cancer Institute |
| NRI | non-responder imputation |
| OC | observed cases |
| PD | pharmacodynamics |
| PK | Pharmacokinetic |
| PPS | per protocol set |
| PT | preferred term |
| RA | rheumatoid arthritis |
| RF | rheumatoid factor |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SDAI | simple disease activity index |
| SI | Système International |
| SJC | swollen joint counts |
| SJC28 | swollen joint counts in 28 joints |
| SJC66 | swollen joint counts in 66 joints |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| TEMAV | treatment-emergent markedly abnormal laboratory value |
| TJC | tender joint counts |
| TJC28 | tender joint counts in 68 joints |
| TJC68 | tender joint counts in 28 joints |
| TLG | tables, listings, and graphs |
| TNF-RI | tumor necrosis factor receptor-I |
| TRACP-5b | tartrate resistant acid phosphatase 5b |

| Abbreviation | Term |
|--------------|-------------------------------------------|
| VAS | visual analog scale |
| VCAM-1 | vascular cell adhesion molecule-1 |
| VEGF | vascular endothelial growth factor |
| WHO DD | World Health Organization Drug Dictionary |

#### 3 INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to describe the procedures and the statistical methods that will be used to analyze and report results for Eisai Protocol E6011-J081-202.

Statistical methods of Treatment Phase is provided in this document. Also, weeks 0 to 12 of the Treatment Phase is defined as Core Treatment Phase, and weeks 0 to 24 of the Treatment Phase is defined as Entire Treatment Phase

## 3.1 Study Objectives

## 3.1.1 Primary Objectives

- To evaluate the efficacy of E6011 by comparing ACR20 response rate at Week 12 with placebo as the primary endpoint
- To evaluate the safety and tolerability of E6011

## 3.1.2 Secondary Objective

• To evaluate the pharmacokinetics (PK) and immunogenicity of E6011

## 3.1.3 Exploratory Objective

• To explore the PK/pharmacodynamics (PD) and biomarkers of E6011

# 3.2 Overall Study Design and Plan

This study is a multicenter, randomized, double-blind, placebo-controlled, parallel-group comparison study. E6011 and placebo groups are set for the study. Subjects will receive E6011 400 mg or placebo at Weeks 0, 1, 2, and every 2 weeks until weeks 10 and then E6011 200 mg or 400 mg every 2 weeks between Weeks 12 and 22.

The study consists of Screening, Observation, Treatment, Extension, and Follow-up Phases.

Undergoing screening assessments within 42 days prior to the study treatment, subjects with the certain eligibility confirmed in the Observation Phase will be allocated into either of the E6011 or placebo group at a 1:1 ratio through dynamic allocation using the following factors: number of biologics with inadequate response, C- reactive protein (CRP) level at Screening

Eisai  FINAL Version 1.0: 4 Jun2018

Phase. Subjects who will continue the study beyond Week 12 will be further randomized to E6011 200 mg or 400 mg administrations at a 1:1 ratio in each group (E6011 or placebo group).

In the Treatment Phase (24 weeks), subjects will receive either E6011 400 mg or placebo at Weeks 0, 1, 2, and every 2 weeks subsequently until Week 10 and then E6011 200 mg or 400 mg every 2 weeks between Weeks 12 and 22 in a double-blind manner.

Subjects who complete evaluations at Week 24 of the Treatment Phase will enter the Extension Phase. The Extension Phase is up to Week 104 from the starting of the study treatment, and subjects will receive an open-label E6011 200 mg every 2 weeks until Week 102. When subjects insufficiently respond to the treatment or when their disease relapses in the Extension Phase (show no improvement from Observation Phase in both of tender joint counts (TJC) and swollen joint counts (SJC) at 2 consecutive assessments with an interval of  $\geq$ 1 week), a dose escalation will be allowed only once (6 administrations of E6011 400 mg every 2 weeks).

Follow-up investigations will be conducted on-site 28 days after the completion of the study or the discontinuation of the treatment, and either an on-site or telephone-interview investigation will be conducted 70 days after the last dosing.

## 4 DETERMINATION OF SAMPLE SIZE

Since the objectives for the study are to explore the efficacy and safety of E6011 repeated subcutaneous administration in RA subjects inadequately responding to biologics, the sample size was not based on statistical considerations. However the sample sizes of 30 for each treatment group will have about 80% power to detect a difference in response rate of 35% if ACR20 response rate of placebo is 20% to 25% based on a chi-square test.

#### 5 STATISTICAL METHODS

All descriptive statistics for continuous variables will be reported using mean, standard deviation (SD), median, minimum and maximum. Categorical variables will be summarized as number (percentage) of subjects.

## 5.1 Study Endpoints

## 5.1.1 Primary Endpoint

• ACR20 response rate at Week 12


The ACR20 response is defined as if the following 3 criteria (ACR components) are met:

- 1. Greater than or equal to 20% reduction from baseline in the TJC in 68 joints (TJC68)
- 2. Greater than or equal to 20% reduction from baseline in the SJC in 66 joints (SJC66)
- 3. Greater than or equal to 20% reduction from baseline in at least 3 of the following 5 assessments:
  - Physician's Global Assessment of Disease Activity (VAS)
  - Patient's Global Assessment of Disease Activity (VAS)
  - Patient's Assessment of Pain (VAS)
  - HAQ-DI
  - CRP

## 5.1.2 Secondary Endpoints

- ACR20, ACR50, and ACR70 response rate at each visit (excluding ACR20 at Week 12)
- Values and change from baseline in ACR components (TJC, SJC, VAS [pain/disease activity assessments by subjects and disease activity assessment by physicians], functional assessment by subjects [HAQ-DI], and CRP·ESR), DAS28-ESR, DAS28-CRP, SDAI, and CDAI at each visit
- EULAR response criteria at each visit; subjects will be classified based on DAS28-ESR and DAS28-CRP
- Remission rates in DAS28-ESR, DAS28-CRP, SDAI, CDAI, and Boolean at each visit The ACR50 response is defined similar to the ACR20 with a 50% reduction.

The ACR70 response is defined similar to the ACR20 with a 70% reduction.

The DAS28-CRP calculates on the following formula, and disease activity is categorized as High at > 4.1, Moderate at > 2.7 and  $\le 4.1$ , Low at  $\le 2.7$ , and Remission at  $\le 2.3$ .

```
0.56 \times sqrt\{TJC \text{ in } 28 \text{ joints } (TJC28)\} + 0.28 \times sqrt\{SJC \text{ in } 28 \text{ joints } (SJC28)\} + 0.36 \times ln\{CRP (mg/dL) \times 10 + 1\} + 0.014 \times - Patient's Global Assessment of Disease Activity (VAS) (mm) + 0.96
```

The DAS28-ESR will be calculated on the following formula, and disease activity is categorized as High at > 5.1, Moderate at > 3.2 and <= 5.1, Low at <= 3.2, and Remission at < 2.6.

 $0.56 \times \text{sqrt}\{\text{TJC28}\} + 0.28 \times \text{sqrt}\{\text{SJC28}\} + 0.70 \times \ln\{\text{ESR (mm/h})\} + 0.014 \times - \text{Patient's Global Assessment of Disease Activity (VAS) (mm)}$ 

Eisai 

#### **EULAR Response Criteria:**

| | DAS28 change from baseline | | |
|---|---|---|---|
| Present DAS28 | <-1.2 | >=-1.2 and $<-0.6$ | >= -0.6 (missing included) |
| Low | Good response | Moderate response | No response |
| Moderate | Moderate response | Moderate response | No response |
| High | Moderate response | No response | No response |

The CDAI will be calculated on the following formula, and disease activity is categorized as High at > 22, Moderate at > 10 and <= 22, Low at <= 10, and Remission at <= 2.8.

- + Patient's Global Assessment of Disease Activity (VAS) (mm) /10
- + Physician's Global Assessment of Disease Activity (VAS) (mm) /10

The SDAI will be calculated on the following formula, and disease activity is categorized as High at > 26, Moderate at > 11 and <= 26, Low at <= 11, and Remission at <= 3.3.

- + Patient's Global Assessment of Disease Activity (VAS) (mm) /10
- + Physician's Global Assessment of Disease Activity (VAS) (mm) /10 + CRP (mg/dL)

The Boolean remission is defined as satisfied all of the following conditions:

- 1.  $TJC68 \le 1$
- 2. SJC66 <= 1
- 3. CRP  $(mg/dL) \leq 1$
- 4. Patient's Global Assessment of Disease Activity (VAS) (mm) <= 10

# 5.2 Study Subjects

## 5.2.1 Definitions of Analysis Sets

Definition of analysis sets are as follows:

- The Full Analysis Set (FAS) is the group of randomized subjects who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement.
- The Full Analysis Set for Entire Treatment Phase (FAS for Entire Treatment Phase) is the group of the re-randomized subjects who received at least 1 dose of study drug after 12 weeks to 24 weeks, and had at least 1 primary efficacy measurement after 12 weeks to 24 weeks.


- The Per Protocol Analysis Set(PPS) is the subset of subjects in the corresponding FAS who do not meet any of following criteria during core treatment phase:
  - Subjects who have any major protocol violations (major inclusion/exclusion violations or other major protocol deviation that affect the evaluation of efficacy
  - ➤ Subjects who are <80% compliant with study drug

A comprehensive list of excluded subjects from the PPS will be verified by the sponsor's medical officer before database lock.

- The Safety Analysis Set is the group of subjects who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
- The Safety Analysis Set for Entire Treatment Phase is the group of the Safety Analysis Set who received study drug after 12 weeks to 24 weeks, re-randomized and had at least 1 safety assessment after 12 weeks to 24 weeks.

The number of subjects randomized, the number and the percentage of subjects included in each analysis set, and the number and the percentage of subjects excluded from each analysis set will be presented by treatment group and overall.

## 5.2.2 Subject Disposition

The numbers of subjects who have provided informed consent, and who are screen failures together with reasons for screening failure will be summarized. The numbers of randomized subjects and the numbers of treated subjects will be summarized for each treatment group and overall. The number and percentage of subjects who completed treatment phase and discontinued the study, and reasons for discontinuation will be summarized for each treatment group and overall.

#### 5.2.3 Protocol Deviations

Major protocol deviation criteria will be established and subjects with major protocol deviations will be identified and documented before the database lock. The protocol deviations identified according to the criteria at study entry and during treatment will not be included in tables, listings, and graphs (TLGs) covered by SAP, but presented in the clinical study report (CSR).

## 5.2.4 Demographic and Other Baseline Characteristics

**Analyses for Core Treatment Phase** 

Demographic and other baseline characteristics for the Safety Analysis Set and FAS will be


summarized for each treatment group (E6011 and placebo) and overall using descriptive statistics.

#### Analyses for Entire Treatment Phase

Demographic and other baseline characteristics for the Safety Analysis Set for Entire Treatment Phase and FAS for Entire Treatment Phase will be summarized for each treatment group (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups) and overall using descriptive statistics.

Continuous demographic and baseline variables include:

- > Age
- ➤ Height (cm)
- ➤ Weight (kg)
- $\triangleright$  BMI (kg/m<sup>2</sup>)
- Disease Duration (years)
- ➤ Dose of MTX (mg/week)
- > Number of Biologics
- > Number of Biologics with Inadequate Response
- > Oral Steroid\*1 (mg/day)
- > ACR Components
- TJC68
- SJC66
- TJC28
- SJC28
- CRP (mg/dL) at Screening
- CRP (mg/dL) at Baseline
- ESR (mm/h) at Baseline
- Physician's Global Assessment of Disease Activity (VAS) (mm)
- Patient's Global Assessment of Disease Activity (VAS) (mm)
- Patient's Assessment of Pain (VAS) (mm)
- HAQ-DI
- ➤ DAS28-CRP
- ➤ DAS28-ESR
- CDAI


- > SDAI
- > Serum Rheumatoid Factor (RF) Concentration (IU/mL)

#### Categorical variables include:

- $\rightarrow$  Age (18<= <35, 35<= <50, 50<= <75)
- Sex (Male, Female)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- Race (White, Black or African American, Japanese, Chinese, Other Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Other)
- $\triangleright$  Disease Duration (< 5 years, >= 5 years)
- Disease Duration (< 1 year, 1 year <= < 5 years, 5 years <= < 10 years, 10 years <= < 15 years, >= 15 years)
- Smoking History (Current, Former, Never)
- Current Medical Conditions (Yes, No)
- Prior use of Biologics (TNF\*2 1/2/3/4/>=5, Non-TNF 1/2/3/4/>=5)
- ➤ Number of Biologics with Inadequate Response(TNF\*2 1/2, Non-TNF 1/2, TNF/Non-TNF 1/2)
- Drug experience of MTX (Yes, No)
- > Dose of MTX (< 6 mg/week, 6 mg/week <= < 12 mg/week, >= 12 mg/week)
- Number of Biologics with Inadequate Response (1, 2)
- $\triangleright$  Drug experience of DMARDs except MTX (Yes 1/2/3/4/>= 5, No)
- Continuation of Steroid
- > Serum RF Concentration (Seropositive High Positive/Low Positive, Seronegative)\*3
- Anti-CCP Antibody (Seropositive High Positive/Low Positive, Seronegative)\*4
- Classification of Global Functional Status in RA
- ➤ DAS28-CRP Category (High: >4.1, Moderate: 2.7 < <= 4.1, Low: <= 2.7)
- ➤ DAS28-ESR Category (High: >5.1, Moderate: 3.2 < <= 5.1, Low: <= 3.2)
- ightharpoonup CDAI (High: > 22, Moderate: 10 < <= 22, Low: <= 10)
- > SDAI (High: > 26, Moderate: 11 < <= 26, Low: <= 11)
- $\triangleright$  CRP level at Screening (< 0.6mg/dL, >= 0.6mg/dL)
- $\triangleright$  CRP level at Baseline (< 0.6mg/dL, >= 0.6mg/dL)
- $\triangleright$  ESR level at Baseline (< 28mm/h, >= 28mm/h)

Eisai 

<sup>\*1</sup> Prednisone-equivalent dose

```
*2 Refer section 8.5 "TNF agent"
```

\*3 Categories of Serum RF Concentration are derives as follows:

```
Seropositive: > 15 (IU/mL)

High Positive: > 45 (IU/mL)

Low Positive: 15 <= <= 45 (IU/mL)
```

Seronegative: <= 15 (IU/mL)

\*4 Categories of Anti-CCP Antibody are derives as follows:

```
Seropositive: >= 4.5 (U/mL)

High Positive: > 13.5 (U/mL)

Low Positive: 4.5 <<= 13.5 (U/mL)

Seronegative: < 4.5 (U/mL)
```

Subject data listings will be provided.

#### MEDICAL HISTORY

A subject data listing will be provided.

#### 5.2.5 Prior and Concomitant Therapy

All investigator terms for medications recorded in the case report form (CRF) will be coded to an 11-digit code using the World Health Organization Drug Dictionary (WHO DD) version (Mar2016 or later). The number (percentage) of subjects who took prior and concomitant medications will be summarized on the FAS by treatment group, Anatomical Therapeutic Chemical (ATC) class, and WHO DD preferred term. Prior medications will be defined as medications that stopped before the first dose of study drug. Concomitant medications will be defined as medications that (1) started before the first dose of study drug and were continuing at the time of the first dose of study drug, or (2) started on or after the date of the first dose of study drug.

#### Analyses for Core Treatment Phase

Prior and concomitant medications for FAS will be summarized for each treatment group (E6011 and placebo).


#### Analyses for Entire Treatment Phase

Concomitant medications for FAS for Entire Treatment Phase will be summarized for each treatment group (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups.

A subject data listing of all medications will be provided.

## 5.2.6 Treatment Compliance

Treatment compliance will be described in section 5.6.1.

## 5.3 Data Analysis General Considerations

## 5.3.1 Pooling of Centers

Subjects from all centers will be pooled for all analyses.

## **5.3.2** Adjustments for Covariates

Determination of covariates are as follows:

- Number of Biologics with Inadequate Response (1, 2)
- CRP Level at Baseline (< 0.6 mg/dL, >= 0.6 mg/dL)

## 5.3.3 Multiple Comparisons/Multiplicity

No multiplicity adjustments are planned.

## 5.3.4 Examination of Subgroups

#### Analyses for Core Treatment Phase

The primary efficacy endpoint, ACR50, and ACR70 will be summarized and analyzed by subgroups defined by section 5.2.4 for categorical variables. Also, forest plot will be created by subgroups for comparison of response rate at primary efficacy endpoint.

Additional subgroup analyses may also be conducted, if deemed appropriate.


#### **Analyses for Entire Treatment Phase**

No subgroup analyses are planned for this study.

## 5.3.5 Handling of Missing Data, Dropouts, and Outliers

For the efficacy analyses, approaches to handling missing data for continuous variables will be the observed cases (OC) method and the last observation carried forward (LOCF) method; binary variables and EULAR response criteria will be the observed cases (OC) method, the last observation carried forward (LOCF) method and the non-responder imputation (NRI) method as each visit.

For the safety analyses and biomarker analyses for continuous value, descriptive statistics are used OC method and LOCF method, this is applied only the last observation of each phase, in tables and figures.

In the cases of laboratory result contains less (or more) than quantitation limit value is treated as:

- a. zero, when less than quantitation limit value,
- b. quantitation limit value, when more than quantitation limit value.

In the cases of pharmacokinetic data, refer "8.2 Convention for Pharmacokinetic data handling".

#### 5.3.6 Other Considerations

## **5.3.6.1** Total number of joints

For the calculation of the total number of joints that are tender/swollen, If any joints are not evaluable, the score is prorated by taking the number of joints that are tender/swollen divided by the number of evaluable joints and multiplied by the target number of joints, rounded to nearest integer. If assessment of joints are "Not Done", the joints will be handled as tender and swollen.

#### **5.3.6.2** HAQ subcategory score

The HAQ-DI is composed of 20 items in 8 categories (Dressing and Grooming, Hygiene, Arising, Reach, Eating, Grip, Walking, Activities). To calculate the HAQ-DI, the highest sub-category score determines the value for each category, there must be responses in at least


6 of the 8 categories or else a HAQ-DI cannot be computed. The category scores are then averaged into an overall HAQ-DI.

HAQ-DI = (Amount of score with all categories) / (Number of categories scored)

## 5.4 Efficacy Analyses

#### Analyses for Core Treatment Phase

The FAS will be used as the primary population for the efficacy analyses, while the PPS will be used as a supportive analysis.

## Analyses for Entire Treatment Phase

The FAS for Entire Treatment Phase will be used as the population for the efficacy analyses

## 5.4.1 Primary Efficacy Analyses

#### Analyses for Core Treatment Phase

ACR20 response rate at Week 12 will be analyzed using a logistic regression model, Number of Biologics with Inadequate Response and CRP Level at Baseline as covariates, for the comparison between placebo and E6011. Significance level is  $\alpha$ =0.025 (one-sided).

Hypothesis for logistic regression model is:

$$\begin{cases} H_0: & \frac{Odds_{400 mg}}{Odds_{Placebo}} = 1 \\ H_1: & \frac{Odds_{400 mg}}{Odds_{Placebo}} > 1 \end{cases}$$

Subjects with missing primary efficacy endpoint due to early discontinuation or other reasons will be considered non-responders. ACR20 response rate and its 2-sided 95% confidence interval of normal approximation for each treatment group will be calculated. The difference in ACR20 response rate between E6011 and placebo and its 2-sided 95% confidence interval of normal approximation will also be calculated.

## 5.4.2 Secondary Efficacy Analyses

#### Analyses for Core Treatment Phase

For ACR20 (excluding Week 12), ACR50, and ACR70, similar analyses as primary analyses


will be conducted. For each component of ACR (TJC, SJC, VAS [pain assessment and disease activity assessment by subjects, and disease activity assessment by physicians], functional assessment by subjects (HAQ-DI) and CRP·ESR), DAS28-ESR, DAS28- CRP, SDAI, and CDAI in each visit, the values and the changes from baseline will be summarized by treatment group(E6011 and placebo). The changes from baseline will also be analyzed using ANCOVA with baseline value, Number of Biologics with Inadequate Response, and CRP Level at Baseline as covariates. The significance level for comparisons between placebo and E6011 is  $\alpha$ =0.05 (2-sided).

For DAS28-ESR and DAS28-CRP, frequency and percentage of each classification (no response, moderate response, good response) by EULAR response criteria will be summarized by treatment group and visit in a shift table. For DAS28-ESR, DAS28-CRP, SDAI and CDAI, frequency and percentage of each category (Remission, Low, Moderate, High) will be summarized by treatment group and visit in a shift table. For remission rates in DAS28-ESR, DAS28-CRP, SDAI, CDAI, and Boolean, similar analyses as primary analyses will be conducted.

The mean of variables (ACR components, DAS28-CRP, DAS28-ESR, CDAI and SDAI) and change from baseline - visit will be displayed by treatment group (E6011 and placebo). ACR response rate - visit, including week 12, will be displayed by treatment group. Bar chart of each variables (ACR response rate, remission rate in DAS28-CRP, DAS28-ESR, CDAI, SDAI and Boolean) will be displayed at week 12. Stacked bar chart of DAS28-CRP and DAS28-ESR by EULAR response criteria will be displayed at week 12. Stacked bar chart of category of DAS28-CRP and DAS28-ESR will be displayed at baseline and week 12.

#### Analyses for Entire Treatment Phase

Each efficacy endpoint for Entire Treatment Phase will be summarized by treatment group (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups) and time point as described below.

For ACR20, ACR50, and ACR70, response rate and its 2-sided 95% confidence interval will be calculated. For each component of ACR (TJC, SJC, VAS [pain assessment and disease activity assessment by subjects, and disease activity assessment by physicians], functional assessment by subjects (HAQ-DI) and CRP·ESR), DAS28-ESR, DAS28- CRP, SDAI, and CDAI, the values and the changes from baseline will be summarized.

For DAS28-ESR and DAS28-CRP, frequency and percentage of each classification (no response, moderate response, good response) by EULAR response criteria will be summarized in a shift table. For DAS28-ESR, DAS28-CRP, SDAI and CDAI, frequency and percentage of each category (Remission, Low, Moderate, High) will be summarized in a shift table. For remission rates in DAS28-ESR, DAS28-CRP, SDAI, CDAI, and Boolean, remission rate and its 2-sided 95% confidence interval will be calculated.

The mean of variables (ACR components, DAS28-CRP, DAS28-ESR, CDAI and SDAI) and


change from baseline - visit will be displayed by treatment group. ACR response rate - visit will be displayed by treatment group. Bar chart of each variables (ACR response rate, remission rate in DAS28-CRP, DAS28-ESR, CDAI, SDAI and Boolean) will be displayed at week 12 and week 24. Stacked bar chart of DAS28-CRP and DAS28-ESR by EULAR response criteria will be displayed at week 12 and week 24. Stacked bar chart of category of DAS28-CRP and DAS28-ESR will be displayed at baseline and week 12 and week 24.

All efficacy endpoints for the treated subjects will be listed.

## 5.4.3 Other Efficacy Analyses

No other efficacy analyses are planned for this study.

# 5.5 Pharmacokinetic, Pharmacodynamic, Pharmacogenomic, and Other Biomarker Analyses

## 5.5.1 Pharmacokinetic Analyses

Serum E6011 Concentration

Serum PK samples for PK analyses will be collected on Week 0 (predose), Week 1 (predose), Week 2 (predose), Week 4 (predose), Week 8 (predose), Week 12 (predose), Week 16 (predose), Week 20 (predose), Week 24 (predose).

#### Analyses for Core Treatment Phase

The Safety Analysis Set will be used for PK analyses.

<Table>

Individual serum concentration values of E6011 will be listed and summarized using descriptive statistics (n, mean, standard deviation, median, minimum and maximum) and nominal time point. The data of time points in subject with interruption will not be included on calculation of summary statistics.

<Figure>

The individual serum E6011 concentration—time profile will be displayed in linear and semilog scales using actual sampling times.


The mean serum concentrations of E6011 will be displayed using nominal blood sampling times with standard deviation in linear and semi-log scales.

#### Analyses for Entire Treatment Phase

The Safety Analysis Set for Entire Treatment Phase will be used for PK analyses.

<Table>

Individual serum concentration values of E6011 from Entire Treatment Phase will be listed and summarized using descriptive statistics (n, mean, standard deviation, median, minimum and maximum) by dose (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups) and nominal time point. The data of time points in subject with interruption will not be included on calculation of summary statistics.

<Figure>

The individual serum E6011 concentration—time profile from Entire Treatment Phase will be displayed in linear and semi—log scales using actual sampling times in the same graph by dose (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups).

The mean serum concentrations of E6011 will be displayed using nominal blood sampling times with standard deviation in linear and semi-log scales by dose in the same graph.

Actual sampling time and serum concentrations of E6011 for each subject will be listed.

# 5.5.2 Pharmacodynamic, Pharmacogenomic, and Other Biomarker Analyses

#### **5.5.2.1** Pharmacodynamic, Pharmacogenomic Analyses

No Pharmacodynamic and Pharmacogenomic analyses are planned for this study.

## 5.5.2.2 Other Biomarker Analyses

#### Analyses for Core Treatment Phase

Biomarker analyses for this period will be performed using the FAS.


Summary statistics for serum RF concentration, serum anti-CCP antibody concentration, and serum matrix metalloproteinase-3 concentration, serum tartrate resistant acid phosphatase 5b (TRACP-5b) concentration, serum cytokine concentration, serum leucine-rich alpha-2 glycoprotein 1 (LRG1) concentration, serum angiopoietin 2 (Ang2) concentration, Vectra<sup>TM</sup> DA and it's component (vascular cell adhesion molecule-1 (VCAM-1), epidermal growth factor (EGF), vascular endothelial growth factor (VEGF)-A, interleukin (IL)-6, tumor necrosis factor receptor-I (TNF-RI), serum matrix metalloproteinase-1, serum matrix metalloproteinase-3, YKL-40, leptin, resistin, SA and CRP) value, change from baseline and percent change from baseline, by treatment group (E6011 and placebo groups) and time point, will be calculated.

## **Analyses for Entire Treatment Phase**

Biomarker analyses for this period will be performed using the FAS for Entire Treatment Phase.

Similar analyses as described in Core Treatment Phase will be conducted by treatment group (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups).

Exploratory investigations of the relationship between efficacy and biomarkers will be conducted. Details and results of analyses of immunocytes such as blood CX3CR1-positive cells in the 400 mg group will be provided in a separate report, and will not be included in the clinical study report. All other biomarkers will be collected on baseline and postbaseline, referring section 8.1.3 "Time window".

Subject data listings will be provided.

#### 5.5.2.3 Immunogenicity Analyses

#### Analyses for Core Treatment Phase

Immunogenicity analyses for this period will be performed using the Safety Analysis Set.

The percentage and frequency of occurrences will be calculated for serum anti-E6011 antibodies and E6011-induced anti-E6011 antibodies by treatment group (E6011 and placebo groups) and time point. If anti-E6011 antibody develops, the frequency and percentage of any anti-E6011 antibody neutralization activity and isotypes will be calculated.


## Analyses for Entire Treatment Phase

Immunogenicity analyses for this period will be performed using the Safety Analysis Set for Entire Treatment Phase.

Similar analyses as described in Core Treatment Phase will be conducted by treatment group (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups).

Subject data listings will be provided.

## 5.6 Safety Analyses

Safety variables include treatment-emergent adverse events (TEAEs), clinical laboratory parameters, vital signs, 12-lead ECG results, chest x-ray, neurological findings, and blood CD4 positive cell count. Day 1 for all safety analyses will be defined as the date of the first dose of study drug.

#### Analyses for Core Treatment Phase

All safety analyses for this period will be performed on the Safety Analysis Set.

Safety data, presented by treatment group (E6011 and placebo groups), will be summarized on an "as treated" basis using descriptive statistics (eg, n, mean, SD, median, minimum, maximum for continuous variables; n [%] for categorical variables).

#### **Analyses for Entire Treatment Phase**

Unless otherwise specified, safety analyses for this period will be performed on the Safety Analysis Set for Entire Treatment Phase. Similar analyses as described in the Core Treatment Phase will be conducted by treatment group (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups).

#### 5.6.1 Extent of Exposure

Analyses for Core Treatment Phase

Eisai 

The extent of exposure to study drug will be characterized by duration of exposure, number of injection and study medication compliance for each treatment group. Definition of analysis items are as follows:

- ➤ Duration of exposure (weeks) = ( Date of Last Dose Date of First Dose + 14 ) / 7
- ➤ Number of Injection = Count of records with non-zero treatment
- ➤ Study Medication Compliance (%) = Number of Injection / Number of Expected Injection \* 100

Analyses for Entire Treatment Phase

Similar analyses as described in Core Treatment Phase will be conducted by treatment group (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups) except duration of study treatment at placebo.

Subject data listings will be provided.

#### 5.6.2 Adverse Events

#### Analyses for Core Treatment Phase

The AE verbatim descriptions (investigator terms from the CRF) will be classified into standardized medical terminology using the Medical Dictionary for Regulatory Activities (MedDRA). Adverse events will be coded to the MedDRA (Version 19.0 or higher) lower level term (LLT) closest to the verbatim term. The linked MedDRA preferred term (PT) and primary system organ class (SOC) are also captured in the database. A treatment-emergent adverse event (TEAE) is defined as an AE that emerges during treatment, having been absent at pretreatment (Baseline) or

- Reemerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or
- Worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.

Only those AEs that are treatment-emergent will be included in summary tables.

A subject will be counted only once within an SOC and PT, even if the subject experienced more than 1 TEAE within a specific SOC and PT.

The TEAEs will be summarized by treatment group and E6011 overall. The incidence of follow TEAEs will be reported as the number (percentage) of subjects with TEAEs by SOC and PT:


- TEAEs
- TEAEs by maximum grade
- Serious TEAEs
- Treatment Related, TEAEs
- Treatment Related, TEAEs by maximum grade
- Treatment Related, Serious TEAEs

## Analyses for Treatment Phase (Weeks 12 to 24)

Similar analyses as described in Core Treatment Phase will be conducted by treatment group (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups).

#### Analyses for Entire Treatment Phase (Weeks 0 to 24)

Similar analyses as described in Core Treatment Phase will be conducted by treatment group (placebo/200 mg, placebo/400 mg, 400 mg/200 mg, and 400 mg/400 mg groups).

When the analyses for this period will be conducted, the incidence of follow TEAEs will also be reported:

- TEAEs leading to study drug withdrawn
- TEAEs leading to interruption of study drug
- TEAEs leading to reduction from study drug
- Treatment Related, TEAEs leading to study drug withdrawn
- Treatment Related, TEAEs leading to interruption of study drug
- Treatment Related, TEAEs leading to reduction from study drug

In the analyses for Core Treatment Phase and Entire Treatment Phase, the AEs emerged until disposition on Week 12/24 are intended, but for patients who discontinued in Treatment Phase, the AEs emerged until 70 days after the last dose are intended

Subject data listings of All AEs, SAEs, AEs leading to death, leading to study drug withdrawn or leading to interruption from study drug will be provided.


## 5.6.3 Laboratory Values

Laboratory results will be summarized using Système International (SI) units. For quantitative parameters listed in protocol Section 9.5.1.5.3, the actual value and the change from baseline to each postbaseline visit will be summarized by visit and treatment group using descriptive statistics. Qualitative parameters listed in protocol Section 9.5.1.5.3 will be summarized using frequencies (number and percentage of subjects), and changes from baseline to each postbaseline visit and to end of treatment will be reported using shift tables. Percentages will be based on the number of subjects with both nonmissing baseline and relevant postbaseline results.

Laboratory test results will be assigned a low/normal/high (LNH) classification according to whether the value was below (L), within (N), or above (H) the laboratory parameter's reference range. Within-treatment comparisons for each laboratory parameter will be based on 3-by-3 tables (shift tables) that compare the baseline LNH classification to the LNH classification at each postbaseline visit and at the end of treatment. Similar shift tables will be used to compare the baseline LNH classification to the LNH classification for the highest and lowest value during the study.

The Sponsor's Grading for Laboratory Values using CTCAE v4.0 presents the criteria that will be used to identify subjects with treatment-emergent markedly abnormal laboratory values (TEMAVs). Except for phosphate, a TEMAV is defined as a postbaseline value with an increase from baseline to a grade of 2 or higher. For phosphate, a TEMAV is defined as a postbaseline value with an increase from baseline to a grade of 3 or higher. When displaying the incidence of TEMAVs, each subject will be counted once in the laboratory parameter high and in the laboratory parameter low categories, as applicable.

Laboratory results versus visit by treatment group will be displayed using box-plot.

Subject data listings of Laboratory test results and TEMAV will be provided.

#### 5.6.4 Vital Signs

Descriptive statistics for vital signs parameters (systolic and diastolic BP, pulse, temperature, and weight) and changes from baseline will be presented by visit and treatment group.

Subject data listings will be provided.

## 5.6.5 Electrocardiograms

Shift tables will be presented changes from baseline in 12-lead ECG interpretation (normal/abnormal, not clinically significant/abnormal, clinically significant) by visit and treatment group.


Subject data listings will be provided.

## 5.6.6 Other Safety Analyses

#### 5.6.6.1 Chest X-Ray

Shift tables will be presented changes from baseline in chest x-ray (normal/abnormal, not clinically significant/abnormal, clinically significant) by visit and treatment group.

Subject data listings will be provided.

#### 5.6.6.2 Neurological findings

Descriptive statistics for neurological findings will be presented by visit and treatment group.

Subject data listings will be provided.

#### 5.6.6.3 Blood CD4 positive cell counts

For Blood CD4 positive cell counts, the actual value and the change from baseline to each postbaseline visit will be summarized by visit and treatment group using descriptive statistics. Blood CD4 positive cell counts will be assigned a low/normal/high (LNH) classification according to whether the value was below (L), within (N), or above (H) the it's reference range. Within-treatment comparisons will be based shift tables that compare the baseline LNH classification to the LNH classification at each postbaseline visit.

Subject data listings will be provided.

## 5.7 Other Analyses

## 5.7.1 Anti-JCV Antibody Test

Anti-JCV antibody test result (positive or negative) is judged according to the results of screen assay and inhibition assay.

Subject data listings will be provided.

Eisai 

## 5.8 Exploratory Analyses

Exploratory analyses may be conducted as appropriate. Any exploratory analyses that are performed will be appropriate titled and labeled as exploratory and will be clearly distinguished from planned analyses when results are reported in the Clinical Study Report.

## 5.9 Extension Phase Analyses

SAP for extension phase will be separately prepared and finalized before database lock.

#### **6 INTERIM ANALYSES**

No interim analyses are planned for this study.

## 7 CHANGES IN THE PLANNED ANALYSES

If the SAP needs to be revised after the study starts, the sponsor will determine how the revision impacts the study and how the revision should be implemented. The details of the revision will be documented and described in the clinical study report.

Deletion in the planned analyses for protocol are as follows:

- Efficacy Analysis
  - The changes from baseline will be summarized using values at Week 12 as baseline.
- Safety Analysis
  - The changes from baseline will be summarized using values at Week 12 as baseline.

Additions in the planned analyses for protocol are as follows:

- Efficacy Analysis
  - ➤ frequency and percentage of each category (Remission, Low, Moderate, High) of DAS28-ESR, DAS28-CRP, CDAI and SDAI will be summarized by treatment group and visit in a shift table.
  - ➤ The mean of variables (ACR components, DAS28-CRP, DAS28-ESR, CDAI and SDAI) and change from baseline visit will be displayed by treatment group.
  - ACR response rate visit, including week 12, will be displayed by treatment group.

Eisai 

- ➤ Bar chart of each variables (ACR response rate, remission rate in DAS28-CRP, DAS28-ESR, CDAI, SDAI and Boolean) will be displayed at week 12 and week 24.
- Stacked bar chart of DAS28-CRP and DAS28-ESR by EULAR response criteria will be displayed at week 12 and week 24.
- Stacked bar chart of category of DAS28-CRP and DAS28-ESR will be displayed at baseline and week 12 and week 24.
- ACR50, ACR70 will be summarized and analyzed by subgroups defined by section 5.2.4 for categorical variables.
- Forest plot will be created by subgroups for comparison of response rate at primary efficacy endpoint.

## • Extent of Exposure

➤ The extent of exposure to study drug will be characterized by number of injection, cumulative dose expected, cumulative dose and study medication compliance for each treatment group.

#### Adverse Events

- The incidence of follow TEAEs will be reported as the number (percentage) of subjects with TEAEs by SOC and PT:
  - ♦ Serious TEAEs
  - → TEAEs leading to discontinuation from study drug
  - ♦ TEAEs leading to interruption of study drug
  - ♦ TEAEs leading to reduction from study drug
  - ♦ Treatment Related, Serious TEAEs
  - ❖ Treatment Related, TEAEs leading to discontinuation from study drug
  - ♦ Treatment Related, TEAEs leading to interruption of study drug
  - → Treatment Related, TEAEs leading to reduction from study drug

#### Laboratory Values

- P Qualitative parameters listed in protocol Section 9.5.1.5.3 will be summarized using frequencies (number and percentage of subjects), and changes from baseline to each postbaseline visit and to end of treatment will be reported using shift tables.
- Percentages will be based on the number of subjects with both nonmissing baseline and relevant postbaseline results.
- Each subject will be counted once in the laboratory parameter high and in the laboratory parameter low categories.


- Laboratory results versus visit by treatment group will be displayed using box-plot.
- Other Analyses
  - Anti-JCV antibody test result listings will be provided.

## 8 DEFINITIONS AND CONVENTIONS FOR DATA HANDLING

## 8.1 Baseline, Time Windows for statistical analyses

#### 8.1.1 Definition of baseline value

The baseline value was defined as the most recent value reported just before first dosing.

## 8.1.2 Definition of change from baseline and percent change from baseline

Change from baseline is defined as postbaseline value minus baseline value. Percent change from baseline is defined as follows:

% Change from baseline = (Change from baseline/Baseline) \* 100

For any Baseline value of 0, the subject's corresponding percent change from baseline will not be included in the summary statistics table.

#### 8.1.3 Time windows

Time windows are defined as Table 8.1 to Table 8.7 for each assessment. Observation that has the most recent date-time on base date-time is adopted if plural observations exist in the time window. Observation recorded later is adopted if they recorded in that same period.

Table 8.1 Definition of time windows and calculated visits for vital signs and Serum E6011 concentration

| Visit | Base date | Time windows |
|---|---|---|
| Week 1 (Day 8) | Date of first drug<br>administration + 7 days | Base date - 3 days <= < Base date + 3 days |
| Week 2 (Day 15) | Date of first drug<br>administration + 14 days | Base date - 4 days <= < Base date + 7 days |
| Week 4 (Day 29) | Date of first drug<br>administration + 28 days | Base date - 7 days <= < Base date + 14 days |

Eisai 

| Visit | Base date | Time windows |
|---|---|---|
| Week 8 - Week 24<br>by 4 weeks | Date-time of first drug<br>administration + X * 7<br>days (Week X) | Base date - 14 days <= < Base date + 14 days |

Table 8.2 Definition of time windows and calculated visits for Physical findings, administration site finding

| Visit | Base date | Time windows |
|---|---|---|
| Week 1 (Day 8) | Date of first drug<br>administration + 7 days | Base date - 3 days <= < Base date + 3 days |
| Week 2 (Day 15) | Date of first drug<br>administration + 14 days | Base date - 4 days <= < Base date + 7 days |
| Week 4 (Day 29) | Date-time of first drug<br>administration + 28 days | Base date - 7 days <= < Base date + 14 days |
| Week 8 - Week 12<br>by 4 weeks | Date-time of first drug<br>administration + X * 7<br>days (Week X) | Base date - 14 days <= < Base date + 14 days |
| Week 24 | Date-time of first drug<br>administration + 168<br>days | Base date - 14 days <= < Base date + 14 days |

Table 8.3 Definition of time windows and calculated visits for Joint assessment, ESR, VAS, HAQ, Laboratory tests (include Hematology, blood chemistry, urinalysis, RF, anti-CCP antibody and matrix metalloproteinase-3)

| Visit | Base date | Time windows |
|---|---|---|
| Week 2 (Day 15) | Date of first drug<br>administration + 14 days | Base date - 4 days <= < Base date + 7 days |
| Week 4 (Day 29) | Date-time of first drug<br>administration + 28 days | Base date - 7 days <= < Base date + 14 days |
| Week 8 - Week 24<br>by 4 weeks | Date-time of first drug<br>administration + X * 7<br>days (Week X) | Base date - 14 days <= < Base date + 14 days |

Table 8.4 Definition of time windows and calculated visits for body weight, 12-lead ECG, Chest x-ray, Pregnancy test, Neurological findings, Blood CD4 positive cells, Autoantibody,


Serum KL-6,  $\beta$  D glucan, Vasculitis marker tests, Serum TRACP-5b concentration, Vectra  $^{\text{TM}}$  DA

| Visit | Base date | Time windows |
|---|---|---|
| Week 12 - Week<br>24 by 12 weeks | Date-time of first drug<br>administration + X * 7<br>days (Week X) | Base date - 14 days <= < Base date + 14 days |

Table 8.5 Definition of time windows and calculated visits for Serum anti-E6011 antibody

| Visit | Base date | Time windows |
|---|---|---|
| Week 4 (Day 29) | Date-time of first drug<br>administration + 28 days | Base date - 7 days <= < Base date + 14 days |
| Week 8 - Week 24 by 4 weeks | Date-time of first drug<br>administration + X * 7<br>days (Week X) | Base date - 14 days <= < Base date + 14 days |

Table 8.6 Definition of time windows and calculated visits for Serum cytokine concentration, LRG1, Ang2

| Visit | Base date | Time windows |
|---|---|---|
| Week 4 (Day 29) | Date-time of first drug<br>administration + 28 days | Base date - 7 days <= < Base date + 14 days |
| Week 12 - Week<br>24 by 12 weeks | Date-time of first drug<br>administration + X * 7<br>days (Week X) | Base date - 14 days <= < Base date + 14 days |

Table 8.7 Definition of time windows and calculated visits for Anti-JCV antibody test

| Visit | Base date | Time windows |
|---|---|---|
| Week 24 | Date-time of first drug<br>administration + 168<br>days | Base date - 14 days <= < Base date + 14 days |

# 8.2 Pharmacokinetic data handling

## 8.2.1 Lower Limit of Quantification of E6011 Serum Concentration

The LLOQ of E6011 serum concentration is 0.1 µg/mL.


## 8.2.2 BLQ Handling for Developing Concentration-Time Profiles

When developing individual concentration-time profiles, BLQ values will be handled according to 302-104.00-MNL for non-compartmental pharmacokinetic analysis.

## 8.2.3 BLQ Handling for Developing Tables

When developing tables, BLQ values will be handled according to 302-104.00-MNL for non-compartmental pharmacokinetic analysis.

## 8.2.4 Handling of anomalous concentration values

Handling anomalous concentration values will follow the 302-104.00-MNL for non-compartmental pharmacokinetic analysis.

## 8.2.5 General Rules for Presentation of Drug Concentrations

When presenting individual/raw (raw, hereafter) values and summary statistics, the following rule will be applied: for drug concentrations, all summary statistics (mean, median, geometric mean, standard deviation (SD) and coefficient variation (CV)) will have 3 significant digits.

## 8.3 Imputation rule for partial date

#### 8.3.1 Date of Diagnosis

Imputation rule for date of diagnosis is as follows:

- Complete date: Date as reported on CRF.
- Year and Month are not missing but Day is missing: Year and Month as reported on CRF, Date as 15th
- Year is not missing but Month and Day are missing: Year as reported on CRF, Month and Day as July 1st.
- Year is missing or Date is completely missing: Missing


#### 8.3.2 Medication

Imputation rule for medication start date is as follows:

- Complete date: Date as reported on CRF
- Year and Month are not missing but Day is missing: Year and Month as reported on CRF, Day as 1st
- Year is not missing but Month and Day are missing: Year as reported on CRF, Month and Day as January 1st
- Year is missing or Start Date is completely missing: Missing

Imputation rule for medication end date is as follows:

- Complete date: Date as reported on CRF
- Year and Month are not missing but Day is missing: Date of death or Year and Month as reported on CRF, last day of the reported month, which is earlier
- Year is not missing but Month and Day are missing: Year as reported on CRF, Month and Day as December 31st
- Year is missing or Start Date is completely missing: Missing

#### 8.3.3 Adverse Events

Imputation rule for adverse event start date is as follows:

- Year and Month are not missing but Day is missing
  - Year and Month are the same as year and month of the earliest among non-missing values of first dosing date of study Treatment and imputed AE end date: The earliest among non-missing values of first dosing date of study Treatment and imputed AE end date
  - Year and Month are not the same as year and month of the earliest among nonmissing values of first dosing date of study Treatment and imputed AE end date: Year and Month as reported on CRF, Day as 1st
- Year is not missing but Month and Day are missing
  - Year is the same as year of the earliest among non-missing values of first dosing date of study Treatment and imputed AE end date: The earliest among non-missing values of first dosing date of study Treatment and imputed AE end date
  - Year is not the same as year of the earliest among non-missing values of first dosing date of study Treatment and imputed AE end date: Year as reported on CRF, Month and Day as January 1st


Completely missing: First dosing date or imputed AE end date, which is earlier

Imputation rule for adverse event end date is as follows:

- Outcome is 'fatal' and End Date is not complete date: Date of death
- Outcome is 'fatal' and End Date is complete date
  - > different from the date of death: Comfirm to CDM
  - > same as the date of death: Date of death
- Outcome is not 'fatal' and date of death is not missing
  - Year and Month are the same as the year and month of date of death: Date of death
  - Year and Month are not the same as the year and month of date of death: Year and Month as reported on CRF, Day as the last day of the month
  - Year is the same as the year of date of death: Date of death
  - Year is not the same as the year of date of death: Year as reported on CRF, Month and Day as December 31st
  - > Completely missing: Date of death
- Outcome is not 'fatal' and date of death is missing
  - Year and Month are not missing but Day is missing: Year and Month as reported on CRF, Day as the last of month
  - ➤ Year is not missing but Month and Day are missing, and Year is before the Year of date of discontinuation from study: Year as reported on CRF, Month and Day as December 31st
  - Year is not missing but Month and Day are missing, and Year is same as the Year of date of discontinuation from study: Date of discontinuation from study
- Outcome is marked 'Recovered' or 'Recovered with sequelae': Date of discontinuation from study
- Outcome is missing or is 'Not recovered', 'Recovering' or 'Unknown', or Year is missing or Start Date is completely missing: Missing
- Year, Month and Day are all missing and date of death is not missing: Date of death

## 8.4 Decimal places

Decimal places (DP) for descriptive statistics, except PK analysis, is defined as follows:

• Mean: Significant digits + 1

• SD: Significant digits + 2


- Median: Significant digits + 1
- Min, Max: Significant digits
- Percentage of frequency: fixed one decimal place

DP for the derived parameter is defined as follows:

Mean: fixed 3 DP
SD: fixed 4 DP
Median: fixed 3 DP
Min, Max: fixed 2 DP

DP for the other calculated result is defined as follows:

- Confidence Interval: fixed 2 DP
- Pvalue: fixed 4 DP, except < 0.0001. When < 0.0001, as is.

Summary of change from baseline is based on significant digits of each parameter, and percent change from baseline is defined as 1 DP.

## 8.5 TNF Agent

Medications as TNF agent are extracted at ATC4 Code = L04AB.

#### 9 PROGRAMMING SPECIFICATIONS

The rules for programming derivations and dataset specifications are provided in separate documents.

#### 10 STATISTICAL SOFTWARE

All statistical analyses will be performed using SAS version 9.3 or later.

# 11 MOCK TABLES, LISTINGS, AND GRAPHS

The study TLG shells will be provided in a separate document, which will show the content and format of all tables, listings, and graphs in detail.


# 12 REFERENCES

Not Applicable.

Eisai 

Statistical Analysis Plan E6011-J081-202

## 13 APPENDICES

# 13.1 National Institute for Health: Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

National Cancer Institute (NCI) CTCAE version 4.0 May 2009 is available online at:

https://evs.nci.nih.gov/ftp1/CTCAE/Archive/CTCAE\_4.0\_2009-05-29\_QuickReference\_5x7.pdf

CTCAE grades for selected laboratory parameters are listed in the table below, where ULN is the upper limit of normal and LLN is the lower limit of normal.

| | NCI Common Terminology Criteria for Adverse Events (CTCAE) - SI Units | | | | |
|---|---|---|---|---|---|
| Lab Parameter | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Hematology | | | | | |
| Hemoglobin (low) | < LLN - 100 (g/L) | < 100 - 80 (g/L) | < 80 - 65 (g/L) | | Death |
| Hemoglobin (high) | Increase in $> 0$ - 20 (g/L) | Increase in $>20 - 40 \text{ (g/L)}$ | Increase in $> 40$ (g/L) | | |
| | above ULN or above | above ULN or above | above ULN or above | | |
| | baseline if baseline is | baseline if baseline is | baseline if baseline is | | |
| | above ULN | above ULN | above ULN | | |
| Platelet Count (PLT) (low) | < LLN - 75.0 (10^9/L) | < 75.0 - 50.0 (10^9/L) | < 50.0 - 25.0 (10^9/L) | < 25.0 (10^9/L) | |
| White Blood Cell Count | < LLN - 3.0 (10^9/L) | < 3.0 - 2.0 (10^9/L) | < 2.0 - 1.0 (10^9/L) | < 1.0 (10^9/L) | |
| (WBC) (low) | | | | | |
| White Blood Cell Count | | | > 100 (10^9/L) | | Death |
| (WBC) (high) | | | | | |
| Lymphocytes (low) | < LLN - 0.8 (10^9/L) | < 0.8 - 0.5 (10^9/L) | < 0.5 - 0.2 (10^9/L) | < 0.2 (10^9/L) | |
| Lymphocytes (high) | | > 4 - 20 (10^9/L) | > 20 (10^9/L) | | |
| Neutrophils (low) | < LLN - 1.5 (10^9/L) | < 1.5 - 1 (10^9/L) | < 1 - 0.5 (10^9/L) | < 0.5 (10^9/L) | |
| Blood Chemistry | | | | | |
| Albumin (low) | < LLN - 3 (g/dL); | < 3 - 2 (g/dL); | < LLN - 2 (g/dL); | | Death |
| | < LLN - 30 (g/L) | < 30 - 20 (g/L) | < 20 (g/L) | | |
| Alkaline Phosphatase (high) | > ULN - 3.0 x ULN | > 3.0 - 5.0 x ULN | > 5.0 - 20.0 x ULN | > 20.0 x ULN | |
| Alanine Aminotransferase | > ULN - 3.0 x ULN | > 3.0 - 5.0 x ULN | > 5.0 - 20.0 x ULN | > 20.0 x ULN | |
| (high) | | | | | |
| Amylase (high) | > ULN - 1.5 x ULN | > 1.5 - 2.0 x ULN | > 2.0 - 5.0 x ULN | > 5.0 x ULN | |

Eisai 

FINAL Version 1.0: dd JUL 2017

Statistical Analysis Plan E6011-J081-202

| | NCI Common Terminology Criteria for Adverse Events (CTCAE) - SI Units | | | | |
|---|---|---|---|---|---|
| Lab Parameter | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| Aspartate Aminotransferase | > ULN - 3.0 x ULN | > 3.0 - 5.0 x ULN | > 5.0 - 20.0 x ULN | > 20.0 x ULN | |
| (high) | | | | | |
| Total Bilirubin (high) | > ULN – 1.5 x ULN | > 1.5 - 3.0 x ULN | > 3.0 - 10.0 x ULN | > 10.0 x ULN | |
| Corrected Calcium*, serum- | < LLN - 2.0 (mmol/L); | < 2 - 1.75 (mmol/L); | < 1.75 - 1.5 (mmol/L); | < 1.5 (mmol/L); | Death |
| low (hypocalcemia) | < LLN - 8.0 (mg/dL) | < 8.0 - 7.0 (mg/dL) | < 7.0 - 6.0 (mg/dL) | < 6.0 (mg/dL) | |
| Corrected Calcium*, serum- | > ULN – 2.9 (mmol/L); | > 2.9 - 3.1 (mmol/L); | > 3.1 - 3.4 (mmol/L); | > 3.4 (mmol/L); | Death |
| high (hypercalcemia) | > ULN – 11.5 (mg/dL) | > 11.5 – 12.5 (mg/dL) | > 12.5 - 13.5 (mg/dL) | > 13.5 (mg/dL) | |
| Cholesterol (high) | > ULN - 300 (mg/dL); | > 300 - 400 (mg/dL); | > 400 - 500 (mg/dL); | > 500 (mg/dL); | |
| | > ULN - 7.75 (mmol/L) | > 7.75 - 10.34 (mmol/L) | > 10.34 - 12.92 (mmol/L) | > 12.92 (mmol/L) | |
| Creatinine (high) | > 1 - 1.5 x baseline; | > 1.5 - 3.0 x baseline; | > 3.0 x baseline; | > 6.0 x ULN | |
| | > ULN - 1.5 x ULN | > 1.5 - 3.0 x ULN | > 3.0 - 6.0 x ULN | | |
| Gammaglutamyltransferase | > ULN - 3.0 x ULN | > 3.0 - 5.0 x ULN | > 5.0 - 20.0 x ULN | > 20.0 x ULN | |
| (high) | | | | | |
| Glucose, serum-low | < LLN - 55 (mg/dL); | <55 - 40 (mg/dL); | < 40 - 30 mg/dL; | < 30 mg/dL; | Death |
| (hypoglycemia) | < LLN - 3.0 (mmol/L) | <3.0 - 2.2 (mmol/L) | < 2.2 - 1.7 mmol/L | < 1.7 mmol/L | |
| Glucose, serum-high | > ULN - 160 (mg/dL); | > 160 - 250 (mg/dL); | > 250 - 500 (mg/dL); | > 500 (mg/dL); | Death |
| (hyperglycemia) | > ULN - 8.9 (mmol/L) | > 8.9 - 13.9 (mmol/L) | > 13.9 - 27.8 (mmol/L) | > 27.8 (mmol/L) | |
| Phosphate, serum-low | <lln -="" 2.5="" dl;<="" mg="" td=""><td>&lt;2.5 - 2.0 mg/dL;</td><td>&lt;2.0 - 1.0 mg/dL;</td><td>&lt;1.0 mg/dL;</td><td>Death</td></lln> | <2.5 - 2.0 mg/dL; | <2.0 - 1.0 mg/dL; | <1.0 mg/dL; | Death |
| (hypophosphatemia) | <lln -="" 0.8="" l<="" mmol="" td=""><td>&lt;0.8 - 0.6 mmol/L</td><td>&lt;0.6 - 0.3 mmol/L</td><td>&lt;0.3 mmol/L;</td><td></td></lln> | <0.8 - 0.6 mmol/L | <0.6 - 0.3 mmol/L | <0.3 mmol/L; | |
| Potassium, serum-low | <lln -="" 3.0="" l<="" mmol="" td=""><td></td><td>&lt;3.0 - 2.5 mmol/L</td><td>&lt;2.5 mmol/L</td><td>Death</td></lln> | | <3.0 - 2.5 mmol/L | <2.5 mmol/L | Death |
| (hypokalemia) | | | | | |
| Potassium, serum-high | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L | >7.0 mmol/L | Death |
| (hyperkalemia) | | | | | |
| Sodium (Hyponatremia) (low) | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L;</td><td>Death</td></lln> | - | <130 - 120 mmol/L | <120 mmol/L; | Death |
| Sodium (Hypernatremia) | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L | >160 mmol/L; | Death |
| (high) | | | | | |
| Triglyceride | 150 - 300 (mg/dL); | > 300 - 500 (mg/dL); | > 500 - 1000 (mg/dL); | > 1000 (mg/dL); | Death |
| (hypertriglyceridemia) (high) | 1.71 - 3.42 (mmol/L) | > 3.42 - 5.7 (mmol/L) | > 5.7 - 11.4 (mmol/L) | > 11.4 (mmol/L) | |
| Uric Acid (hyperuricemia) | > ULN - 10 (mg/dL); | - | | > 10 (mg/dL); | Death |
| (high) | <= 0.59 (mmol/L) | | | > 0.59 (mmol/L) | |
| Urinalysis | | | | | |
| Protein | 1+ | 2+ or higher | | | |
| Other | | | | | |
| Blood CD4 Positive Cell | < LLN - 0.5 (10^9/L) | < 0.5 - 0.2 (10^9/L) | < 0.2 - 0.05 (10^9/L) | < 0.05 (10^9/L) | |
| Counts | , , , | | | | |

<sup>\*</sup> Corrected serum calcium by albumin should be referred. If serum albumin is <4.0~g/dL, the corrected calcium will be calculated using the following formula:

 $Corrected\ calcium\ (mg/dL) = Total\ calcium\ (mg/dL) - 0.8\ x\ [Albumin\ (g/dL) - 4]$ 

Eisai 

FINAL Version 1.0: dd JUL 2017

Statistical Analysis Plan E6011-J081-202

As to Alkaline Phosphatase and  $\gamma$ -GTP, criteria for Grade 2 is changed from ULN x 2.5 (in the CTCAE) to ULN x 3.0.

# 13.2 Sponsor's Grading for Determining Markedly Abnormal Laboratory Results

Except for phosphate, a TEMAV is defined as a postbaseline value with an increase from baseline to a grade of 2 or higher. For phosphate, a TEMAV is defined as a postbaseline value with an increase from baseline to a grade of 3 or higher.

Eisai 

# SIGNATURE PAGE



Eisai 

FINAL Version 1.0: 4 JUN 2018